CLINICAL TRIAL: NCT01804907
Title: Feasibility of Non-pharmacological Insomnia Therapy in People Living With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00032846
Record Dates: First submitted 2013-03-04; First posted 2013-03-05 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Insomnia; Sleep Efficiency
Keywords: HAART adherence; HIV; Fatigue; treatment
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Fatigue | interventions — Cognitive Behavioral Therapy; Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT (Experimental): Cognitive Behavioral Therapy
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Behavioral Modification (Sham Comparator): Standard sleep hygiene education/desensitization therapy
  Interventions: Behavioral: Behavioral Modification

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy
  Arms: CBT
Behavioral: Behavioral Modification
  Arms: Behavioral Modification

SUMMARY:
To establish with a prospective randomized placebo-controlled study the feasibility of allied-health personnel-administered cognitive behavioral insomnia therapy (CBTI) as a means of improving HIV/AIDS treatment adherence.

ELIGIBILITY:
Inclusion Criteria:

* provide documentation of HIV seropositivity, and have been on current HAART (Highly Active AntiRetroviral Therapy) or antiretroviral regimen without any foreseeable reason to discontinue the HAART during the course of the study;
* males or females age 18-75 years of age;
* ≥3 month history of insomnia meeting standard psychiatric criteria for insomnia based on DSISD;
* sleep onset latency (SOL) and/or wake after sleep onset (WASO) greater than 30 minutes, with a corresponding sleep time of less than 6.5 hours at least 3 nights per week (as measured by the 7-day sleep diary);
* be able to read, understand, and sign an informed consent form before entering into the study and must be willing to comply with all study procedures as well as to agree to participate for the entire study period.

Exclusion Criteria:

* use of any medication with a significant effect on sleep/wake function within 5 half-lives of baseline or during the study including hypnotics, over-the-counter sleep aides, sedating antidepressants or sedating anxiolytics;
* history or DSISD (Duke Insomnia Sleep Diagnostics) suggests sleep disorder other than insomnia (e.g., sleep apnea, narcolepsy, periodic leg movements, etc.), or have insomnia associated with circadian rhythm disturbances, such as night or rotating shift work or travel across more than four time zones in the 14 days before Initial Screening (Visit 1) or during the study;
* clinically significant unstable medical or psychiatric condition, or have any clinically significant abnormal finding in physical examination, neurological assessment, or vital signs, as determined by the Investigator;
* self reports typical consumption of more than five alcoholic beverages on a single day or greater than 14 alcoholic beverages weekly at Initial Screening (Visit 1);
* have used any investigational drug within 30 days or five half-lives (whichever is longer) prior to Initial Screening (Visit 1), or plans to use an investigational drug during the study;
* unable to give informed consent or comply with study procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Sleep Efficiency | Week 1, 2,3, and 4
  Patients evaluated weekly for change in sleep efficiency.

SECONDARY OUTCOMES:
Adherence to HAART | Week 1, 2,3, and 4
  Evaluated once weekly for changes in medication adherence.
Fatigue | Week 1, 2,3, and 4
  Changes in reported fatigue levels measured weekly, via the Paper Fatigue Scale (PFS), and the HIV-Related Fatigue Scale (HRFS).

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States